CLINICAL TRIAL: NCT06859073
Title: A Phase 1, Double-blinded, Placebo-controlled Study of Single Ascending Doses of NNC4004-0002 in Adults With Asymptomatic Hyperuricemia
Brief Title: A Research Study to Evaluate the Safety of NNC4004-0002 When Given to Participants With Asymptomatic Hyperuricemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NN4004-8071; U1111-1317-9961 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC4004-0002 (Experimental): Participants will receive a single dose of NNC4004-0002 injected subcutaneously. Trial will include up to 6 ascending single-dose cohorts.
  Interventions: Drug: NNC4004-0002
- Placebo (Placebo Comparator): Participants in each cohort will receive placebo matched to NNC4004-0002 injected subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC4004-0002 — NNC4004-0002 will be given as a single ascending dose via subcutaneous route.
  Arms: NNC4004-0002
Drug: Placebo — Placebo matched to NNC4004-0002 will be given via subcutaneous route.
  Arms: Placebo

SUMMARY:
This study will evaluate an investigational drug called NNC4004-0002. "Investigational" means NNC4004-0002 has not been approved for sale/ for clinical use or for the use described in this study/ by any regulatory authority. Its use in this study is experimental. This will be the first time that NNC4004-0002 will be given to human. This study will be testing the ability of the study medicine to lower serum uric acid. The main aim of this study will be to see if the new study medicine is safe and tolerated by the body after a single dose of study medicine in adults with asymptomatic hyperuricemia. Participants will either get NNC4004-0002 (the study medicine), or saline. Which treatment the participant get will be decided by chance. The participant will get the medicine as an injection under their skin. Depending on the dose they will receive, participant may need more than one injection. The study will last for about 19 months in total. The participant will take part in the study for about 7 months. Participant will have approximately 14 visits to the clinic and one of them will be a 4 night in-house stay.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 35 to 75 years of age at the time of signing the informed consent form (ICF).
* Considered to be generally healthy based on medical history, physical examination, and the re-sults of vital signs, electrocardiogram, and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Body mass index (BMI) 20 to 35 kilogram per meter square (kg/m2) (both inclusive) at screening.
* Serum uric acid levels greater than or equal to (≥) 6.8 miligram per decileter (mg/dL) to less than or equal (≤) 12 mg/dL on 2 consecutive screening samples (the first at the screening visit [V1], and the second taken at V2 [day -1]; samples at least 7 days apart).

Exclusion Criteria:

* Female who is pregnant, breastfeeding, or intends to become pregnant or is of childbearing po-tential and not using an adequate contraceptive method.
* Male of reproductive age who, or whose female partner(s), is not using an adequate contraceptive method.
* Present or prior history of gout, or present or prior use of serum Uric acid (sUA) lowering medication.
* Serious cardiovascular or hepatic disease, current or past malignancies, or chronic debilitating neurologic, gastrointestinal, or inflammatory diseases.
* History or current diagnosis of chronic history kidney disease.
* Screening alanine transaminase (ALT) or aspartate aminotransferase (AST) values greater than (>) 2 multiply by (×) upper limit normal (ULN) or total bilirubin >1.5× ULN.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-emergent adverse event (TEAEs) | From dosing (day 1) until end of study (approximately 28 weeks)
  Count

SECONDARY OUTCOMES:
AUC(0-72): The area under the NNC4004-0002 plasma concentration-time curve from time zero to the 72 hours after a single dose | From dosing (day 1) to 72 hours postdose
  microgram•hour/mililiter (μg•h/mL)
Cmax: The maximum concentration of NNC4004-0002 in plasma | From dosing (day 1) to 72 hours postdose
  microgram/mililiter
tmax: The time from dose administration to the maximum plasma concentration of NNC4004-0002 | From dosing (day 1) to 72 hours postdose
  Hours
Renal clearance | From time of dose to 72 hours postdose
  Liter/hour (L/h)
Changes in serum Uric Acid (sUA) over time | From baseline through the end of the study (approximately 28 weeks)
  miligram/deciliter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - PAREXEL Glendale/LA EPCU, Glendale, California
  - PAREXEL Intl - EPCU-Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: https://novonordisk-trials.com